CLINICAL TRIAL: NCT06524349
Title: Utilization of a 3D Printed Customized Knee Extender and At-Home Rehabilitation Program on Patient Outcomes Following ACL Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SH AOSSM Grant Study
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Tear; Anterior Cruciate Ligament Rupture
Keywords: 3D printing; knee extender device
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Study team member who obtains knee measurements will be blinded to study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D printed knee extender device (Experimental): Participants will utilize a 3D printed knee extender device and an at-home home rehabilitation program designed to be used with the 3D printed knee extender device.
  Interventions: Device: 3D printed knee extender device
- Standard Rehabilitation (No Intervention)

INTERVENTIONS:
Device: 3D printed knee extender device — Participants will receive a 3D printed knee extender device with sealed water bottles and an at-home rehabilitation program designed to be used with the 3D printed knee extender device.
  Arms: 3D printed knee extender device

SUMMARY:
The purpose of this study is to explore patient outcomes associated with, the use of a 3D printed knee extender device, in conjunction with an at-home rehabilitation program, for patients who are performing knee rehabilitation after anterior cruciate ligament (ACL) surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a primary ACL rupture. Secondary knee pathology such as, but not limited to bone edema, strains, and meniscal pathology are acceptable as long as the primary injury and indication for surgery is the ACL rupture.
* Able and willing to adhere to the study procedures
* Able to consent for self-, or able to assent for self with parental consent

Exclusion Criteria:

* Pregnancy
* Non-English speaking

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Extension Range of Motion | Change from baseline range of motion to 6 week post-ACL surgery follow up visit.
  Knee extension range of motion is measured by a trained study member who is blinded to the participant's study group using a goniometer. Participants are seated on the exam table with their leg maximally extended. The center of the goniometer is placed over the lateral epicondyle of the affected knee. One of the goniometer arms is aimed proximally, pointing toward the greater trochanter of the hip. The other arm is aimed distally, pointing toward the lateral malleolus of the ankle. The study member then reads the angle created by the arms of the goniometer in this position.
Time to Achieve Full Knee Extension | Through study completion, an average of 6 weeks.
  Full knee extension will be measured at home by participants by placing a clicking device under their knee which will produce an audible "click" when the knee is fully extended, and the clicker is depressed. Participants in the control and experimental groups will notify the study team during weekly follow up surveys whether they are able to depress the clicker or not.

SECONDARY OUTCOMES:
Knee Swelling | through study completion, an average of 6 weeks.
  Participants knee swelling is measured by a trained study member who is blinded to the participant's study group. Circumference of the knee is used as a proxy for knee swelling, and is measured by wrapping a tape measure around the circumference of the knee just proximal to the superior pole of the patella with resting tension.
Average Daily Pain Level | From baseline until their 6-week post-ACL surgery follow up visit, an average of 6 weeks.
  Participants will complete a weekly follow up survey which will ask them about their average pain level.
Water bottles used with knee extender device | From baseline until their 6-week post-ACL surgery follow up visit, an average of 6 weeks.
  Participant in the experimental arm will provide the average number of water bottles used to weigh down their knee sling during their weekly follow up survey.
Minutes Spent Using Knee Extender Device | From baseline until their 6-week post-ACL surgery follow up visit, an average of 6 weeks.
  Participants in the experimental arm will provide the average number of minutes spend using their knee extender device during their weekly follow up survey

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Skelley, MD, Principal Investigator — Sanford Health
Locations (2):
- United States (2):
  - Sanford Orthopedics and Sports Medicine, Fargo, North Dakota
  - Sanford Orthopedics and Sports Medicine, Sioux Falls, South Dakota